CLINICAL TRIAL: NCT04278378
Title: Blood Pressure Lowering Effect of B-vitamins in Adults With a Genetic Pre-disposition to Elevated Blood Pressure.
Acronym: RAFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REC/11/0081
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Blood Pressure
Keywords: Blood pressure; Central hemodynamics; Methylenetetrahydrofolate reductase (MTHFR); Folate polymorphism; Riboflavin; Folic acid
MeSH Terms: interventions — Riboflavin; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Riboflavin (Active Comparator): 1.6 mg riboflavin / day for 24 weeks
  Interventions: Dietary Supplement: Riboflavin
- Folic Acid (Experimental): 0.4 mg folic acid/ day for 24 weeks
  Interventions: Dietary Supplement: Folic acid
- Riboflavin + Folic Acid (Experimental): 1.6mg Riboflavin + 0.4 mg Folic Acid / day for 24 weeks
  Interventions: Dietary Supplement: Riboflavin; Dietary Supplement: Folic acid
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Riboflavin — 1.6 mg riboflavin / day for 24 weeks
  Arms: Riboflavin; Riboflavin + Folic Acid
Dietary Supplement: Folic acid — 0.4 mg folic acid / day for 24 weeks
  Arms: Folic Acid; Riboflavin + Folic Acid
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Approximately 12% of the world's population have a have a common C677T polymorphism in the gene encoding the folate metabolising enzyme, methylenetetrahydrofolate reductase (MTHFR). Homozygosity for the polymorphism (TT genotype) causes an increased requirement for the B-vitamins folic acid and riboflavin and more importantly results in an increased risk of developing high blood pressure (BP). Previous work from our Centre has demonstrated significantly higher BP in those with the TT genotype. This work has been conducted in cohorts with premature cardiovascular disease (CVD) and hypertension without overt CVD, but the effect in younger, healthier individuals is unexplored. To date our studies have also focused on BP as the primary outcome, but newer markers of vascular health including central pressure and hemodynamics have emerged as superior prognostic indicators of CVD. The effect of the TT genotype on these measures is an area for investigation and may help us understand the mechanism linking the genotype with BP, which is currently unknown. As adults with the TT genotype have increased requirements for riboflavin and folic acid, and BP in TT adults appears to be riboflavin dependent, the influence of these vitamins on central measures is an area for consideration. Study Design This is an observational study investigating the blood pressure profiles of healthy adults aged 18-65 years, stratified by MTHFR genotype. Apparently healthy adults will be recruited from workplaces and the general community across Northern Ireland and screened for the polymorphism via buccal swab. Those with the TT genotype and a similar number of non-TT (i.e. CC/CT) genotype individuals will be contacted and asked to come to a one-off appointment. Brachial BP will be assessed by an electronic BP monitor, central BP and central haemodynamics (augmentation index, augmentation pressure and pulse wave velocity) will be assessed by SphygmoCor XCEL. In addition, anthropometric measurements, health and lifestyle infromation and a blood sample will be obtained. Data will be statistically analysed using SPSS software to if determine differences between gentoype groups exist.

ELIGIBILITY:
Inclusion Criteria:

* MTHFR 677TT genotype, aged at least 18 years old

Exclusion Criteria:

* Taking supplements containing B-vitamins
* Pregnant or planning to conceive
* Taking medications interfering with folate metabolism
* Renal or gastrointestinal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2564 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Change from baseline to 24 weeks
  Office blood pressure

SECONDARY OUTCOMES:
Central blood pressure | Change from baseline to 24 weeks
  Measured using SphygmoCor device
Pulse wave analysis | Change from baseline to 24 weeks
  Measured using SphygmoCor device
Pulse wave velocity | Change from baseline to 24 weeks
  Measured using SphygmoCor device
Red blood cell riboflavin | Change from baseline to 24 weeks
  Measured using erythrocyte glutathione reductase activity coefficient (EGRAC)
Red blood cell folate | Change from baseline to 24 weeks
  Measured by microbiological assay
Serum homocysteine | Change from baseline to 24 weeks
  Measured using an immunoassay
Plasma vitamin B6 | Change from baseline to 24 weeks
  Measured by High Performance Liquid Chromatography

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No